CLINICAL TRIAL: NCT01640418
Title: Prevention of Sacral Pressure Ulcers With Preventive Dressings
Acronym: SACRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL40299.068.12
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Grade I to Grade IV Pressure Ulcers in Higher Risk Patients
Keywords: pressure ulcer; dressing; prevention; higher risk patients
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepilex® Border Sacrum dressings (Experimental): Mepilex® Border Sacrum dressings
  Interventions: Device: Mepilex® Border Sacrum dressings
- Standard Care (No Intervention): Standard Care

INTERVENTIONS:
Device: Mepilex® Border Sacrum dressings — Mepilex® Border Sacrum dressings
  Arms: Mepilex® Border Sacrum dressings

SUMMARY:
In this study we would like to find a way to prevent sacral pressure ulcers in high-risk patients by the use of a Mepilex sacral dressing. The research question we would like to answer is the following: Is the Mepilex sacral dressing a cost-effective dressing for the prevention of grade I to grade IV pressure ulcers in the sacral region in higher-risk hospitalized patients?

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years
* Admission in one of the ten high-risk departments of the azM
* Suspected hospital stay of 5 days or more after admission
* Braden score 19 or less

Exclusion Criteria:

* Age: <18 years
* Pre-existing sacral pressure ulcer
* Pre-existing trauma to the sacrum
* Patient is unable to speak Dutch
* Patients with an inability to give informed consent
* Patients who are unable to give informed consent within 24h after admission
* Patients who are unable to give informed consent before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To compare the number of patients who develop sacral pressure ulcers between the group with the Mepilex® Border Sacrum dressings (Group A) and the group without any sacral dressings (Group B). | 8 weeks
  till hospital release, max 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Bouvy, Principal Investigator — Academic Hospital of Maastricht
Locations (1):
- Academic Hospital of Maastricht, Maastricht, Netherlands